CLINICAL TRIAL: NCT00756080
Title: "Effects of Oral Citrulline on Protein Metabolism in Healthy Humans: a Prospective, Randomized, Double-blind , Cross-over Study"
Brief Title: "Effects of Oral Citrulline on Protein Metabolism in Healthy Humans: a Prospective, Randomized, Double-blind , Cross-over Study" (Citrugrêle)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Dominique DARMAUN, Nantes University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BRD 07/12-D
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2009-01

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): After receiving a 7-day oral supplementation with citrulline, each subject will be admitted to the Clinical Investigation Unit for a half day, after an overnight fast,and will receive a 5-h intravenous infusion of L-[1-13C]leucine (i.e.; leucine labeled with 13C, a stable isotope of carbon) from 8 am to 1 pm. At regular intervals throughout the isotope infusion, blood will be obtained to measure 13C-enrichment in plasma a-keto-isocaproate, the keto acid of leucine, using gas chromatography-mas spectrometry. Simultaneously, 13C-enrichment will be measured in aliquots of expired air CO2 using isotope ratio mass spectrometry, and total CO2 production (VCO2) will be measured using direct calorimetry, respectively. The subject will then leave the hospital, take no treatment for13 days (wash-out period). The study will then be repeated a second time in an identical fashion, after a second 7-day period of oral supplementation with placebo, as a cross-over study design will be used.
  Interventions: Drug: citrulline
- 2 (Placebo Comparator): After receiving a 7-day oral supplementation with placebo, each subject will be admitted to the Clinical Investigation Unit for a half day, after an overnight fast,and will receive a 5-h intravenous infusion of L-[1-13C]leucine (i.e.; leucine labeled with 13C, a stable isotope of carbon) from 8 am to 1 pm. At regular intervals throughout the isotope infusion, blood will be obtained to measure 13C-enrichment in plasma a-keto-isocaproate, the keto acid of leucine, using gas chromatography-mas spectrometry. Simultaneously, 13C-enrichment will be measured in aliquots of expired air CO2 using isotope ratio mass spectrometry, and total CO2 production (VCO2) will be measured using direct calorimetry, respectively. The subject will then leave the hospital, take no treatment for13 days (wash-out period). The study will then be repeated a second time in an identical fashion, after a second 7-day period of oral supplementation with citrulline, as a cross-over study design will be used.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: citrulline — 0.06 G/kg three times/day during 7 days
  Arms: 1
Drug: placebo — placebo (equimolar mixture of 6 non essential amino acids: alanine, aspartate, glycine, histidine, proline, serine) 0,006 g/kg 3 times/day during 7 days
  Arms: 2

SUMMARY:
The specific aim of this study is to determine whether oral citrulline administration enhances whole body protein synthesis in healthy humans in the postabsorptive state. Protein metabolism will be assessed using an intravenous infusion of stable isotope labeled leucine. The investigators hypothesize that citrulline supplementation will decrease leucine oxidation without altering proteolysis, and consequently stimulate protein synthesis .

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult between 18 and 45 years of age
* Absence of any earlier supplementation with citrulline, glutamine, ornithine a-ketoglutarate, or stimol®
* Absence of any treatment with anabolic agents during the month prior to inclusion in the study- No current artificial feeding (enteral or parenteral)
* No renal, cardiac, respiratory or hepatic insufficiency
* No chronic inflammatory disease (intestinal or other
* No current corticotherapy
* Fasting blood glucose below 6mmol/L (126 mg/dL)
* Body mass index between 19 and 24.9
* Patient able to understand benefits and risks of protocol
* Not pregnant, taking oral contraceptive measure if able to procreate
* Subject affiliated to French health insurance (Sécurité Sociale)
* Informed consent form signed
* No concomitant participation to another clinical trial, and compliance with the exclusion period required by law

Exclusion Criteria:

* Subject not fulfilling inclusion criteria
* Subject mentioned in articles L1121-5 to L1121-8 of "code de la santé publique"
* Subject for whom the participation in this clinical trial would result, by cumulating stipends received for other clinical trials, in earning more than 4500 € within 12 consecutive months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To determine whether oral citrulline administration enhances whole body protein synthesis in healthy humans in the psotabsorptive state, as measured using an intravenous infusion of stable isotope labeled leucine

SECONDARY OUTCOMES:
Using a 12-h urine collection, to confirm the positive effect of oral citrulline administration on nitrogen balance observed in preliminary studies (Rougé et al, Am J Physiol 293:G1061, 2007)
To determine whether the putative protein anabolic effect of citrulline is mediated by insulin or insulin-like-growth factor 1 (IGF-1), based on measurement of their plasma concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Darmaun, Professor, Principal Investigator — Nantes University Hospital; Ronan THIBAULD, Doctor, Study Chair — Nantes University Hospital
Locations (1):
- CHU Nantes, Nantes, France